CLINICAL TRIAL: NCT05062330
Title: The TRANQUILITY 2 Trial: Multi-Center Randomized, Double-Masked, Parallel Design, Vehicle-Controlled Phase 3 Clinical Trial to Assess the Efficacy and Safety of 0.25% Reproxalap Ophthalmic Solution Compared to Vehicle in Subjects With Dry Eye Disease
Brief Title: The TRANQUILITY 2 Trial: A Phase 3 Clinical Trial to Assess the Efficacy and Safety in Subjects With Dry Eye Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aldeyra Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADX-102-DED-023
Record Dates: First submitted 2021-09-13; First posted 2021-09-30 (Actual); Results first posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2021-09

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Reproxalap Ophthalmic Solution (0.25%) administered 7 times over two consecutive days (Experimental)
  Interventions: Drug: Reproxalap Ophthalmic Solution (0.25%)
- Vehicle Ophthalmic Solution administered 7 times over two consecutive days (Placebo Comparator)
  Interventions: Drug: Vehicle Ophthalmic Solution

INTERVENTIONS:
Drug: Reproxalap Ophthalmic Solution (0.25%) — Reproxalap Ophthalmic Solution (0.25%) administered 7 times over two consecutive days
  Arms: Reproxalap Ophthalmic Solution (0.25%) administered 7 times over two consecutive days
Drug: Vehicle Ophthalmic Solution — Vehicle Ophthalmic Solution administered 7 times over two consecutive days
  Arms: Vehicle Ophthalmic Solution administered 7 times over two consecutive days

SUMMARY:
The TRANQUILITY 2 Trial: Multi-Center Randomized, Double-Masked, Parallel Design, Vehicle-Controlled Phase 3 Clinical Trial to Assess the Efficacy and Safety of 0.25% Reproxalap Ophthalmic Solution Compared to Vehicle in Subjects with Dry Eye Disease

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age (either gender and any race);
* Reported history of dry eye for at least 6 months prior to Visit 1;
* Reported history of use or desire to use eye drops for dry eye symptoms within 6 months of Visit 1

Exclusion Criteria:

* Clinically significant slit lamp findings at Visit 1 that may include active blepharitis, meibomian gland dysfunction (MGD), lid margin inflammation, or active ocular allergies that require therapeutic treatment, and/or in the opinion of the investigator may interfere with study parameters;
* Diagnosis of an ongoing ocular infection (bacterial, viral, or fungal), or active ocular inflammation at Visit 1;
* Contact lens use within 7 days of Visit 1 or anticipate using contact lenses during the trial;
* Eye drop use within 2 hours of Visit 1;
* Previous laser-assisted in situ keratomileusis (LASIK) surgery within the last 12 months;
* Cyclosporine 0.05% or 0.09% or lifitegrast 5.0% ophthalmic solution use within 90 days of Visit 1;
* Be receiving systemic corticosteroid therapy (not including inhaled corticosteroids) within 14 days of Visit 1 or anticipate such therapy throughout the study period;
* Planned ocular and/or lid surgeries over the study period or any ocular surgery within 6 months of Visit 1;
* Temporary punctal plugs during the study that have not been stable within 30 days of Visit 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 2021-08-28 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2022-03-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Andover Eye Associates (Raynham), Raynham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Reproxalap: Reproxalap ophthalmic solution (0.25%) was administered 7 times over two consecutive days.
- Vehicle: Vehicle ophthalmic solution was administered 7 times over two consecutive days.
Period: Overall Study
Arm/Group | Reproxalap | Vehicle
Started | 181 | 180
Completed | 168 | 168
Not Completed | 13 | 12

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population
Groups:
- Total: Total of all reporting groups
Arm/Group | Reproxalap | Vehicle | Total
Number analyzed (Participants) | 181 | 180 | 361
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 83 | 98 | 181
  >=65 years | 98 | 82 | 180
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (12.2) | 61.9 (12.9) | 63.1 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 126 | 249
  Male | 58 | 54 | 112
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 3 | 13
  Not Hispanic or Latino | 171 | 177 | 348
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 9 | 10 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 25 | 36 | 61
  White | 147 | 132 | 279
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Schirmer Test Mean Change From Baseline
Description: Change from baseline comparison of reproxalap to vehicle for Schirmer test (0 to 35 mm). Higher scores represent greater tear production. The least squares mean (standard error) was derived from a mixed model repeated measures analysis of change from baseline, with baseline as a covariate, and time point and treatment group as factors.
Time Frame: The efficacy assessment period was before and after the final dose on Day 1 (Dose 4). Baseline was approximately two weeks before dosing at Screening.
Population: Intent-to-treat population with observed data only
Measure: Least Squares Mean (Standard Error); unit: length in millimeters
Arm/Group | Reproxalap | Vehicle
Number analyzed (Participants) | 181 | 180
length in millimeters | 1.8 (0.4) | -0.5 (0.4)

2. Primary Outcome: Number of Subject Eyes That Are Schirmer Test Responders
Description: Comparison of reproxalap to vehicle for number of subject eyes that are Schirmer test responders (10 millimeters or more increase from baseline). A generalized estimating equation analysis was performed with baseline as a covariate, and time point and treatment group as factors.
Time Frame: as for outcome 1
Population: Intent-to-treat population with observed data only
Measure: Number; unit: eyes
Arm/Group | Reproxalap | Vehicle
Number analyzed (Participants) | 181 | 180
eyes | 116 | 54
Statistical Analysis 1: Comparison: Reproxalap vs Vehicle; Test type: Superiority; p < 0.0001, Generalized estimating equation; Odds Ratio (OR) = 2.63, 95% CI 2-sided [1.67 to 4.13]

ADVERSE EVENTS:
Time Frame: The safety assessment period was two days.
Arm/Group | Reproxalap | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/181 | 0/180
Serious Adverse Events (participants affected / at risk) | 0/181 | 0/180
Other Adverse Events (participants affected / at risk) | 145/181 | 6/180
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reproxalap (N=181) | Vehicle (N=180)
General disorders and administration site conditions (General disorders) | 145 (145) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-18): https://cdn.clinicaltrials.gov/large-docs/30/NCT05062330/Prot_SAP_000.pdf